CLINICAL TRIAL: NCT06653595
Title: Randomized Control Trial to Evaluate a Breastfeeding Support and Promotion Program to Improve the Health of Premature Babies (PAP-LM)
Brief Title: Breastfeeding Support and Promotion Program to Improve the Health of Premature Babies (PAP-LM)
Acronym: PAP-LM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Mireia Pascual Tutusaus, Principal Investigator, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HCB/2021/0595
Record Dates: First submitted 2024-06-05; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Prematurity; Extreme; Prematurity
Keywords: IBCLC; advance practice nurse; best practice; breastfeeding rates; breastfeeding outcomes; interventions
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: We will be use the random.org program to randomize families into two groups: experimental group (which will receive the intervention) and control group (which will receive usual care).The experimental group intervention will include: 1 pre-discharge face-to-face session, 8 home sessions until 4 months, and 3 telephone sessions until the baby is 6 months old. All sessions will be conducted by an Advanced Practice Nurse and IBCLC Expert in breastfeeding issues.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP (No Intervention): The Control Group receives the usual intervention from the health center, that consists in breastfeeding support in the NICU 1 time/week until hospital discharge.
- EXPERIMENTAL GROUP (Experimental): The Experimental Group receives the PAP-LM programme.
  Interventions: Other: Programme to Support Breastfeeding

INTERVENTIONS:
Other: Programme to Support Breastfeeding — The intervention consists of active support for breastfeeding by a lactation expert and IBCLC until the premature baby is 6 months old. The intervention includes: 1 face-to-face pre-discharge session, 8 home sessions up to 4 months and 3 telephone sessions up to 6 months.
  Arms: EXPERIMENTAL GROUP

SUMMARY:
This study evaluates the effectiveness of a breastfeeding support and promotion program to increase exclusive breastfeeding rates in the preterm group. The intervention is performed by an Advanced Practice Nurse and International Board Certified Breastfeeding Consultant (IBCLC), with high expertise in breastfeeding problems. It is a combination of face-to-face, home care and telephone attention to improve the adherence to breastfeeding. The intervention lasts 6 months.

DETAILED DESCRIPTION:
Will be included moderately premature infants to the Neonatal Unit of the Hospital Clínic who achieve with the inclusion criteria of the study. The sample calculation includes 162 subjects to increase breastfeeding rates to 70% at discharge, 50% at 3 months and 40% at 6 months of the babies. Mothers who wish to exclusively breastfeed up to 6 months and sign the informed consent, will be randomized into the experimental group or control group. The control group will receive usual care and the experimental group will receive 1 pre-discharge face-to-face session, 8 home care sessions up to 4 months and 3 telephone follow-up sessions up to 6 months of baby.

ELIGIBILITY:
Inclusion Criteria:

* Moderate premature
* Late premature babies
* Admitted to the NICU of Hospital Clínic
* Single pregnancy
* Families residing in the Barcelona Metropolitan Area (AMB)
* Families with a good mental health
* Families with a desire for Exclusive Breastfeeding up to 6 months

Exclusion Criteria:

* Maternal diseases that contraindicate breastfeeding
* Mothers with a history of breast surgery
* Mothers with a history of severe hypogalactia
* Premature babies with severe complications
* Premature babies diagnosed with severe CIR

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
BREASTFEEDING RATES | 15 days postpartum, at 3 months and at 6 months postpartum
  Exclusive Breastfeeding or Parcial Breastfeeding

SECONDARY OUTCOMES:
PREMATURE GROWTH | 15 days postpartum, at 3 and 6 months postpartum
  Kilograms, percentiles and Z-scores of weight
PREMATURE HEIGHT | 15 days postpartum, at 3 and 6 months postpartum
  Meters, percentiles and Z-scores of height
PREMATURE CRANIAL PERIMETER | 15 days postpartum, at 3 and 6 months postpartum
  Meters, percentiles and Z-scores of head circumference
PUNTUATION IN DEVELOPMENT WITH ASQ-3 | At 6 months postpartum
  Total puntuation in Ages And Stages Questionnarie of Development (ASQ-3)
MOTHER EFFICACY WITH BREASTFEEDING (USING BSES) | 15 days postpartum and at 6 months postpartum
  The Breastfeeding Self-Efficacy Scale (BSES) is a tool that helps assess how confident a mother feels about her ability to breastfeed. Based on the idea that believing in yourself impacts success, the scale uses 14 questions to measure a mother's sense of capability in different breastfeeding tasks. The higher her score, the more confident she feels. This scale is commonly used by healthcare providers and researchers to better understand where mothers might need extra support, as confidence plays a key role in how long and how successfully they continue breastfeeding.

CONTACTS AND LOCATIONS:
Overall Officials: MIREIA PASCUAL, Principal Investigator — HOSPITAL CLÍNIC I PROVINICIAL DE BARCELONA
Locations (2):
- Spain (2):
  - Rosselló 230, Barcelona
  - C/Sabino de Arana, 1, Barcelona

IPD SHARING:
Plan to Share IPD: No
The information will be confidential. Participation in the study will be voluntary and optional. Participants may leave the study at any time. No data or results will be transferred to patients.

REFERENCES:
- [Background] Bonuck KA, Trombley M, Freeman K, McKee D. Randomized, controlled trial of a prenatal and postnatal lactation consultant intervention on duration and intensity of breastfeeding up to 12 months. Pediatrics. 2005 Dec;116(6):1413-26. doi: 10.1542/peds.2005-0435. PMID 16322166
- [Background] Bonuck K, Stuebe A, Barnett J, Labbok MH, Fletcher J, Bernstein PS. Effect of primary care intervention on breastfeeding duration and intensity. Am J Public Health. 2014 Feb;104 Suppl 1(Suppl 1):S119-27. doi: 10.2105/AJPH.2013.301360. Epub 2013 Dec 19. PMID 24354834
- [Background] Dias de Oliveira L, Justo Giugliani ER, Cordova do Espirito Santo L, Meirelles Nunes L. Counselling sessions increased duration of exclusive breastfeeding: a randomized clinical trial with adolescent mothers and grandmothers. Nutr J. 2014 Jul 17;13:73. doi: 10.1186/1475-2891-13-73. PMID 25033743
- [Background] Gross RS, Mendelsohn AL, Gross MB, Scheinmann R, Messito MJ. Randomized Controlled Trial of a Primary Care-Based Child Obesity Prevention Intervention on Infant Feeding Practices. J Pediatr. 2016 Jul;174:171-177.e2. doi: 10.1016/j.jpeds.2016.03.060. Epub 2016 Apr 21. PMID 27113376
- [Background] Hopkinson J, Konefal Gallagher M. Assignment to a hospital-based breastfeeding clinic and exclusive breastfeeding among immigrant Hispanic mothers: a randomized, controlled trial. J Hum Lact. 2009 Aug;25(3):287-96. doi: 10.1177/0890334409335482. Epub 2009 May 12. PMID 19436060
- [Background] Kools EJ, Thijs C, Kester AD, van den Brandt PA, de Vries H. A breast-feeding promotion and support program a randomized trial in The Netherlands. Prev Med. 2005 Jan;40(1):60-70. doi: 10.1016/j.ypmed.2004.05.013. PMID 15530582
- [Background] Nabulsi M, Tamim H, Shamsedine L, Charafeddine L, Yehya N, Kabakian-Khasholian T, Masri S, Nasser F, Ayash S, Ghanem D. A multi-component intervention to support breastfeeding in Lebanon: A randomized clinical trial. PLoS One. 2019 Jun 14;14(6):e0218467. doi: 10.1371/journal.pone.0218467. eCollection 2019. PMID 31199849
- [Background] O'Reilly SL, McNestry C, McGuinness D, Killeen SL, Mehegan J, Coughlan B, O'Brien EC, O'Brien D, Szafranska M, Brosnan M, Sheehy L, Murtagh R, O'Hagan L, Corbett M, Walsh M, Keogh R, Power P, Woodcock M, Phelan M, Carroll A, Murray S, Scallan C, Dunn E, McAuliffe FM. Multicomponent perinatal breastfeeding support in women with BMI >25: The Latch On multi-centre randomised trial. BJOG. 2024 Aug;131(9):1197-1206. doi: 10.1111/1471-0528.17782. Epub 2024 Feb 12. PMID 38344894
- [Background] Petrova A, Ayers C, Stechna S, Gerling JA, Mehta R. Effectiveness of exclusive breastfeeding promotion in low-income mothers: a randomized controlled study. Breastfeed Med. 2009 Jun;4(2):63-9. doi: 10.1089/bfm.2008.0126. PMID 19239405
- [Background] Tahir NM, Al-Sadat N. Does telephone lactation counselling improve breastfeeding practices? A randomised controlled trial. Int J Nurs Stud. 2013 Jan;50(1):16-25. doi: 10.1016/j.ijnurstu.2012.09.006. Epub 2012 Oct 17. PMID 23084438
- [Background] You H, Lei A, Xiang J, Wang Y, Luo B, Hu J. Effects of breastfeeding education based on the self-efficacy theory on women with gestational diabetes mellitus: A CONSORT-compliant randomized controlled trial. Medicine (Baltimore). 2020 Apr;99(16):e19643. doi: 10.1097/MD.0000000000019643. PMID 32311936